CLINICAL TRIAL: NCT04117269
Title: Clinical Efficacy of an External Shoe Lift in the Contralateral Limb to Improve Healing and Adherence in Patients With Diabetic Foot Ulcers
Brief Title: External Shoe Lift to Improve Healing and Adherence in Patients With Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Raúl Juan Molines Barroso, Phd, Clinical Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/337-E
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Foot Ulcer; Peripheral Neuropathy; Treatment Adherence and Compliance
MeSH Terms: conditions — Diabetic Foot; Peripheral Nervous System Diseases; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External shoe lift (Experimental): Those patients allocated in the experimental group will be supplemented with a external shoe lift in the contralateral limb in their conventional shoes to compensate the differences with the affected foot (using a offloading device to active ulcer).
  Interventions: Device: External shoe lift
- Standard of care (No Intervention): Those patients allocated in the control group will not be supplemented, they will be treated with a standard of care treatment.

INTERVENTIONS:
Device: External shoe lift — Height compensation will be made with cork or EVA (polyurethane + Ethylene Vinyl Acetate) depending the characteristics of the shoe. It will be made by the same orthophaedic technician. The prescription of the heigh of the lift will be made with the patient in a barefoot standing position, a calibre will be used to mark the femoro-tibial joint in both lower limbs in order to rule out the asymmetry. After this, the patient will shod the offloading device in the ulcerated feet and their conventional footwear in the other foot (with the use of their own foot orthosis). 5 millimeters splints will be added under the non affected footwear until the previous mark in both limbs been balanced. The difference in the heigh between limbs will be assessed measuring all the splints used previously
  Arms: External shoe lift

SUMMARY:
Previous researches hipothesize that imposed limb-length discrepancies may discourage adherence in patients with active diabetic foot ulcer and using offloading devices. Our hipothesis is that the use of an external shoe lift contralaterally to the affected foot may improve adherence to offloading devices and improve healing.

ELIGIBILITY:
Inclusion Criteria:

* Plantar diabetic foot ulcer.
* Wagner I and II classification.
* Ulcer area between 1-30 cm square centimeters.
* HbA1c values in the last three months below 11%
* Ankle brachial Index (ABI) value > 0.5.

Exclusion Criteria:

* Diagnosis of Critical Limb Ischaemia definid by TASCC II guideline.
* Presence of foot ulcer in both feet.
* Presence of soft tissue infection.
* Osteomyelitis suspicion.
* Peripheral neuropathy due to different causes than diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of diabetic foot ulcers healed | 12 weeks
  Evaluated by the same clinicians, defined as 100% of epithelialization in absence of exudate

SECONDARY OUTCOMES:
Percentage of diabetic foot ulcers healed | 20 weeks
  Evaluated by the same clinicians, defined as 100% of epithelialization in absence of exudate
Adherence to offloading device | 3 days
  Two pedometer will be used (one inside the vendaje and the other into the offloading device)
Time to healing | 30 weeks
  Time in weeks of diabetic foot ulcer healing

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetic foot Unit Complutense University, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No